CLINICAL TRIAL: NCT07352267
Title: Diagnostic Value and Safety of Endobronchial Ultrasound-guided Transbronchial Mediastinal Cryobiopsy Versus Transbronchial Needle Aspiration in the Diagnosis of Lymphoma: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DETECTION-LYM
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Mediastinal and Hilar Lymphadenopathy
Keywords: Endobronchial ultrasound; Transbronchial needle aspiration; Transbronchial mediastinal cryobiopsy; Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endobronchial ultrasound-guided transbronchial needle aspiration (Experimental)
  Interventions: Procedure: Endobronchial ultrasound-guided transbronchial needle aspiration
- Endobronchial ultasound-guided transbronchial mediastinal cryobiopsy (Experimental)
  Interventions: Procedure: Endobronchial ultrasound-guided tranbronchial mediastinal cryobiopsy

INTERVENTIONS:
Procedure: Endobronchial ultrasound-guided transbronchial needle aspiration — After the target lymph nodes are determined and the safety of needle aspiration is ensured, a 19-G needle will be placed in the working channel of the EBUS scope. The tip of the sheath of the needle will be visible on the endobronchial view, and the needle will then be allowed to pierce the airway wall and enter the lymph node using the jabbing technique under direct ultrasound guidance. A 50-mL syringe will be used to collect 20 mL of aspirates, which will be maintained for 20 s. Each lymph node will be sampled five times to optimize the diagnostic yield. Five passes per node are planned. The samples will not be evaluated on site.
  Arms: Endobronchial ultrasound-guided transbronchial needle aspiration
Procedure: Endobronchial ultrasound-guided tranbronchial mediastinal cryobiopsy — After the target lymph node is located (vascular structures will be excluded via the Doppler function), a tunnel will be made between the target lymph node and the airway wall using a 19-G needle. Subsequently, a 1.1-mm cryoprobe (Erbe 20 402-401, ERBE, Tübingen, Germany) will be inserted through the tunnel and positioned within the target lymph node under EBUS monitoring. The distance between the cryoprobe tip and the lymph node edge will be confirmed to be >5 mm in all four directions. Afterward, the probe will be cooled in liquid carbon dioxide for 5-9 s. A total of three passes will be performed.
  Arms: Endobronchial ultasound-guided transbronchial mediastinal cryobiopsy

SUMMARY:
The goal of this clinical trial is to learn which of two minimally invasive procedures is better at safely diagnosing lymphoma in the mediastinum (chest) in adults (aged 18 and older) who are suspected to have either a new or a returning (relapsed) lymphoma. The main questions it aims to answer are:

Which procedure, endobronchial ultrasound-guided transbronchial mediastinal cryobiopsy (EBUS-TBMC) or endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA), has a higher success rate in obtaining a definitive diagnosis? Is one procedure safer than the other in terms of complications? Researchers will compare the EBUS-TBMC group to the EBUS-TBNA group to see if the cryobiopsy technique leads to better diagnostic results and has a similar or better safety profile.

Participants will:

Be randomly assigned to undergo one of the two diagnostic procedures (EBUS-TBMC or EBUS-TBNA) during a single bronchoscopy session.

Have their tissue samples analyzed by pathologists. Be followed clinically for at least 6 months to confirm the final diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Presence of mediastinal lymphadenopathy of unknown etiology.
* Clinical suspicion of lymphoma, based on any of the following:

Previous history of lymphoma (suspected relapse). Presence of lymphoma at another site. Clinical and radiographic findings suggestive of new isolated mediastinal lymphoma (e.g., isolated idiopathic bulky mediastinal adenopathy with or without systemic symptoms), as assessed by the study bronchoscopists.

Exclusion Criteria:

* A more probable alternative cause for lymphadenopathy is identified (e.g., lung cancer or other non-lymphoproliferative malignancies).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | 7 days after sampling

SECONDARY OUTCOMES:
Diagnostic sensitivity | 7 days after smpling
Incidence of complications | 7 days after sampling
Rate of specimen adequacy | 7 days after sampling